CLINICAL TRIAL: NCT03030365
Title: The Orientation System, the Default-network and Brain Metabolism in Patients With Early Stage Alzheimer's Disease: a Multimodal Functional Study.
Brief Title: Orientation in AD Patients: PET-MR Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, david groshar, Professor, Assuta Medical Center
Other Study IDs: AssutaMC
Record Dates: First submitted 2017-01-08; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Orientation, Disorientation.
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Orientation, Spatial; Confusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Controls: Age matched controls for the various clinical groups will undergo standardly used Magnetic resonance imaging (MRI) protocols, including resting state fMRI, task fMRI, T1 weighted imaging. In addition Patients will receive an intravenous injection of 2-5mCi (millicurie) of 18F (fluorodeoxyglucose) -FDG prior to PET MRI, using "Biograph mMR" PET-MR (3T).
  Interventions: Device: Siemens "Biograph mMR" PET-MR (3T)
- Amnestic Mild cognitive impaired: Patients diagnosed with mild cognitive impairment, exhibiting impairment mostly in memory that is significant but does not interfere with everyday activities.
  Subjects will undergo standardly used Magnetic resonance imaging (MRI) protocols, including resting state fMRI, task fMRI, T1 weighted imaging. In addition Patients will receive an intravenous injection of 2-5mCi of 18F-FDG prior to PET MRI, using "Biograph mMR" PET-MR (3T).
  Interventions: Device: Siemens "Biograph mMR" PET-MR (3T)
- Alzheimer's disease patients: Patients exhibiting significant loss of intellectual ability that interferes with everyday functioning that meet Alzheimer's pattern of decline, and following exclusion of alternative neurodegenerative, cerebrovascular, and metabolic etiologies.
  Subjects will undergo standardly used Magnetic resonance imaging (MRI) protocols, including resting state fMRI, task fMRI, T1 weighted imaging. In addition Patients will receive an intravenous injection of 2-5mCi of 18F-FDG prior to PET MRI, using "Biograph mMR" PET-MR (3T).
  Interventions: Device: Siemens "Biograph mMR" PET-MR (3T)

INTERVENTIONS:
Device: Siemens "Biograph mMR" PET-MR (3T) — Standardly used Magnetic resonance imaging (MRI) protocols, including resting state fMRI, task fMRI, T1 weighted imaging. In addition Patients will receive an intravenous injection of 2-5mCi of 18F-FDG prior to PET MRI.

SUMMARY:
Despite the high prevalence of Alzheimer's disease (AD), its underlying mechanisms remain poorly understood. An emerging body of evidence supports disorientation as an early marker for AD-related neurodegeneration. In this study we intend to collect, coregister and analyze Positron Emission Tomography (PET) and , functional and structural magnetic resonance imaging (MRI, fMRI) data from AD-spectrum patients to establish orientation as core disturbance in AD.

DETAILED DESCRIPTION:
As population aging is progressively contributing to the global burden of dementia, Alzheimer's disease (AD) is gaining recognition as a health-and social-care priority. Evidence converging from recently published works as well as our own preliminary results, propose that orientation is a sensitive marker for preclinical AD-related neurodegeneration.

Our behavioral results show a simple orientation test to surpass currently used neuropsychological tests in classification of patients along the AD spectrum. A subsequential fMRI study revealed the orientation task to preferentially recruit brain regions identified as susceptible to early AD-related cortical atrophy, including the posterior cingulate cortex, parietooccipital sulcus and hippocampus bilaterally, as well as to significantly overlap with the default mode network (DMN) - a set of interconnected brain regions which were independently recognized as highly perturbed in AD.

In an attempt to further support the role of orientation in AD we propose to use co-registration of several modalities of neuroimaging in patients with AD, mild cognitive impairment (MCI) and healthy controls (HC): resting-state fMRI, task-fMRI, structural MRI and co-registered PET.

1. Resting-state functional magnetic resonance (fMRI) imaging detecting temporally synchronous, spatially distributed, spontaneous low frequency blood-oxygen level-dependent signal fluctuations in task-free settings, that are further clustered into maps of functional large-scale neural networks. A major network revealed in rest is the default DMN. DMN includes the posterior cingulate (PCC), inferior parietal (IPL), lateral (LTC) and medial temporal (MTL), and medial prefrontal cortical regions (MPFC), and is known to be involved in self-referential processes including introspection, memory retrieval, daydreaming and orientation.
2. Task fMRI - using this module we recently demonstrated that fMRI activation generated by orientation task in the person, space and time domains activated the PCC, IPL, and MPFC and MTL hubs of the DMN. This task is now to be applied in patients with AD.
3. Structural MRI - a decrease in hippocampus volume is an early imaging finding followed by cortical atrophy as AD progresses.
4. PET - FDG-PET (glucose metabolism) is known to show temporo-parietal hypometabolism in AD.

Considered these findings alongside ongoing research at the dynamics of anatomical and functional AD associated brain dysfunction, we propose a thorough, and to the best of our knowledge, a never before attempted study aimed at linking markers for AD pathology (cortical atrophy, decrease of functional connectivity, cerebral glucose metabolism) to the disruption of specific cognitive faculties, particularly orientation in the space, time and person domains.

ELIGIBILITY:
Inclusion Criteria:

1. subjects aged 50-79 years.
2. patients suffering from memory disorder.
3. Test score mini-mental state examinations higher than 20.

Exclusion Criteria:

1. Contraindication to MR imaging
2. pregnant women.
3. patients with contraindications for injection of gadolinium.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study Population includes patients diagnosed as amnestic mild cognitively impaired, patients suffering from Alzheimer's disease, and age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2019-02-15 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Orientation performance | 1 day
  Evaluation of Performance in orientation task using success rate and response time. Response time and success rate would be combined into an efficacy score: success rate-response time quotient, measured in units of second^-1. A primary effort in this work is to establish a model that links all primary Outcome Measures, in an attempt to examine how pathological markers predict cognitive performance and weather there relations are modulated by fMRI activity.
Cortical atrophy | 1 Day
  Cortical atrophy will be evaluated by applying voxel-based morphometry analysis on T1-weighted images. This outcome would be evaluated as number of voxels significantly different from from a distribution of corresponding voxels gathered from a healthy control cohort. significantly different voxels would be considered atrophic.
Functional connectivity analysis | 1 Day
  Functional connectivity measurements within and between functional networks. This outcome would be evaluated by using correlation values computed between single voxels/region of interest, such that correlation values reflect integrity of functional networks.
Mental-orientation evoked fMRI activity | 1 Day
  Contrasting mental-orientation evoked activity between controls , MCIs and AD. This outcome would be evaluated by applying a contrast between fMRI patterns of activity evoked by the mental-orientation task in clinical groups (AD and MCI) to their control counterparts, to reveal the number and location of voxels showing reduced or increased activity in mental-orientation processing.
[18]F-fluorodeoxyglucose (FDG) uptake | 1 Day
  [18]F-fluorodeoxyglucose glucose analog uptake is measured using positron emission tomography, and is regarded as a marker for neural activity. This outcome would be evaluated by normalizing FDG absorption values and examining voxels statistically different in their metabolic activity relative to highly validated norms.

CONTACTS AND LOCATIONS:
Overall Officials: David Groshar, MD, Principal Investigator — Head of nuclear medicine unit in Assuta Medical Centers

IPD SHARING:
Plan to Share IPD: Undecided
Only in the case where publication of coded data is required\encouraged by the Journal for publication

REFERENCES:
- [Result] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Result] Arzy S, Collette S, Ionta S, Fornari E, Blanke O. Subjective mental time: the functional architecture of projecting the self to past and future. Eur J Neurosci. 2009 Nov;30(10):2009-17. doi: 10.1111/j.1460-9568.2009.06974.x. Epub 2009 Nov 11. PMID 19912333
- [Result] Berrios GE. Disorientation states and psychiatry. Compr Psychiatry. 1982 Sep-Oct;23(5):479-91. doi: 10.1016/0010-440x(82)90161-4. No abstract available. PMID 7140264
- [Result] Buckner RL, Snyder AZ, Shannon BJ, LaRossa G, Sachs R, Fotenos AF, Sheline YI, Klunk WE, Mathis CA, Morris JC, Mintun MA. Molecular, structural, and functional characterization of Alzheimer's disease: evidence for a relationship between default activity, amyloid, and memory. J Neurosci. 2005 Aug 24;25(34):7709-17. doi: 10.1523/JNEUROSCI.2177-05.2005. PMID 16120771
- [Result] deIpolyi AR, Rankin KP, Mucke L, Miller BL, Gorno-Tempini ML. Spatial cognition and the human navigation network in AD and MCI. Neurology. 2007 Sep 4;69(10):986-97. doi: 10.1212/01.wnl.0000271376.19515.c6. PMID 17785667
- [Result] Jheng SS, Pai MC. Cognitive map in patients with mild Alzheimer's disease: a computer-generated arena study. Behav Brain Res. 2009 Jun 8;200(1):42-7. doi: 10.1016/j.bbr.2008.12.029. Epub 2008 Dec 31. PMID 19162077
- [Result] Kunz L, Schroder TN, Lee H, Montag C, Lachmann B, Sariyska R, Reuter M, Stirnberg R, Stocker T, Messing-Floeter PC, Fell J, Doeller CF, Axmacher N. Reduced grid-cell-like representations in adults at genetic risk for Alzheimer's disease. Science. 2015 Oct 23;350(6259):430-3. doi: 10.1126/science.aac8128. PMID 26494756
- [Result] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Result] Monacelli AM, Cushman LA, Kavcic V, Duffy CJ. Spatial disorientation in Alzheimer's disease: the remembrance of things passed. Neurology. 2003 Dec 9;61(11):1491-7. doi: 10.1212/wnl.61.11.1491. PMID 14663030
- [Result] Peer M, Salomon R, Goldberg I, Blanke O, Arzy S. Brain system for mental orientation in space, time, and person. Proc Natl Acad Sci U S A. 2015 Sep 1;112(35):11072-7. doi: 10.1073/pnas.1504242112. Epub 2015 Aug 17. PMID 26283353